CLINICAL TRIAL: NCT01131975
Title: Single Dose Two-Way Crossover, Bioequivalence Study of Lamotrigine 25 mg Chewable Tablets With Lamictal 25 mg Chewable Tablets in Healthy Volunteers Under Fed Condition
Brief Title: Bioequivalence Study of Lamotrigine 25 mg Chewable Tablets of Dr.Reddy's Under Fed Condition
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dr. Reddy's Laboratories Limited (Industry)
Responsible Party: M.S. Mohan / Senior Manager, R&D, Dr. Reddy's Laboratories Limited
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: AAI-US-148
Record Dates: First submitted 2010-05-26; First posted 2010-05-27 (Estimated); Last update posted 2010-06-14 (Estimated); Status verified 2010-06

CONDITIONS: Healthy
Keywords: Bioequivalence; Crossover; Lamotrigine (chewable, dispersible)
MeSH Terms: interventions — Lamotrigine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lamotrigine (chewable, dispersible) (Experimental): Lamotrigine Tablets (chewable, dispersible),25 mg of Dr. Reddy's Laboratories Limited
  Interventions: Drug: Lamotrigine
- Lamictal (Active Comparator): Lamictal Tablets 25 mg of Glaxo SmithKline
  Interventions: Drug: Lamotrigine

INTERVENTIONS:
Drug: Lamotrigine — Lamotrigine Tablets (chewable, dispersible), 25 mg
  Other Names: Lamictal

SUMMARY:
The purpose of this study is to determine the pharmacokinetics and bioequivalence of Lamotrigine formulations after administration of single doses to non-smoking, healthy males and females under fed conditions

DETAILED DESCRIPTION:
A single-dose, two-way, bioequivalence study in up to 24 normal, non-smoking, healthy males and females will be utilized to evaluate the pharmacokinetics and bioequivalence of Lamotrigine chewable dispersible formulations under fed conditions.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females at least 18 years of age inclusive.
* Informed of the nature of the study and given written informed consent.
* Have a body weight within 15% of the appropriate range as defined in the
* 1983 Metropolitan Life Company tables and weighing at least 100 lbs. (Appendix I and II).

Exclusion Criteria:

* Hypersensitivity to Lamotrigine' (Lamictal®), or similar compounds.
* Any history of a clinical condition which might affect drug absorption, metabolism or excretion.
* Recent history (within 1 year) of mental illness, drug addiction, drug abuse or alcoholism.
* Donation of greater than 500 ml of blood in the past 4 weeks prior to study dosing or difficulty in donating blood.
* Received an investigational drug within the 4 weeks prior to study dosing.
* Currently taking any prescription medication, except oral contraceptives, within the 7 days prior to study dosing or over-the-counter medication within 3 days of study dosing; This prohibition does not include vitamins or herbal preparations taken as nutritional supplements for non-therapeutic indications as judged by the attending physician.
* Tobacco use (>5 cigarettes per day) in the 3 months prior to study dosing.
* If female, the subject is lactating or has a positive pregnancy test at screening and prior to each of the two treatment periods. Females of child bearing potential must use a medically acceptable method of contraception throughout the entire study period and for one week after the study is completed. Medically acceptable methods of contraception that may be used by the subject and/or her partner are: oral contraceptives, progestin injection or implants, condom with spermicide, diaphragm with spermicide, IUD, vaginal spermicidal suppository, surgical sterilization of their partner(s) or abstinence. Females taking oral contraceptives must have taken them consistently for at least three months prior to receiving study medication.

Ages: 18 Years to 41 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2003-01; Primary Completion 2003-02 (Actual); Study Completion 2003-03 (Actual)

PRIMARY OUTCOMES:
Bioequivalence based on Cmax and AUC parameters | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Ralph Scallion E.E, M.D., Principal Investigator — AAIPharma
Locations (1):
- AAI Clinic, Chapel Hill, North Carolina, United States